CLINICAL TRIAL: NCT00956475
Title: Quality of Life in Young Adult Survivors of Hematologic Malignancies
Brief Title: Quality of Life in Younger Leukemia and Lymphoma Survivors
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE11Z08; P30CA043703 (NIH); CASE11Z08 (Other: Case Comprehensive Cancer Center); CASE 11Z08-CC607 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Anxiety Disorder; Cancer Survivor; Fatigue; Leukemia; Long-term Effects Secondary to Cancer Therapy in Adults; Lymphoma; Lymphoproliferative Disorder; Pain; Psychosocial Effects of Cancer and Its Treatment; Small Intestine Cancer
Keywords: anxiety disorder; long-term effects secondary to cancer therapy in adults; fatigue; pain; psychosocial effects of cancer and its treatment; cancer survivor; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult Hodgkin lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II adult Hodgkin lymphoma; stage II adult T-cell leukemia/lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system lymphoma; post-transplant lymphoproliferative disorder; cutaneous B-cell non-Hodgkin lymphoma; small intestine lymphoma
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Leukemia; Lymphoma; Lymphoproliferative Disorders; Pain; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Intraocular Lymphoma | interventions — Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: telephone-based intervention — Patients are assessed in a telephone interview using a brief demographic and clinical data form. Patients then undergo quality-of-life assessment by the Cancer Patient/Cancer Survivor Version questionnaire via telephone.
Other: questionnaire administration — Patients are assessed in a telephone interview using a brief demographic and clinical data form. Patients then undergo quality-of-life assessment by the Cancer Patient/Cancer Survivor Version questionnaire via telephone.
Procedure: assessment of therapy complications — questionnaire via telephone
Procedure: fatigue assessment and management — questionnaire via telephone
Procedure: psychosocial assessment and care — questionnaire via telephone
Procedure: quality-of-life assessment — questionnaire via telephone

SUMMARY:
RATIONALE: Collecting information about the effect of hematologic cancer and its treatment on quality of life may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This phase I trial is studying quality of life in younger leukemia and lymphoma survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To collect preliminary data to determine the extent to which there is impairment in quality of life of young adult survivors of hematologic malignancies.
* To identify the most common areas of concern in these survivors.
* To explore patterns of quality-of-life impairment associated with age, gender, and type of treatment (transplant vs non-transplant) in these survivors.

OUTLINE: Patients are assessed in a telephone interview using a brief demographic and clinical data form. Patients then undergo quality-of-life assessment by the Cancer Patient/Cancer Survivor Version questionnaire via telephone.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Survivors of leukemia (i.e., acute myelogenous leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, or chronic lymphocytic leukemia) or lymphoma (i.e., non-Hodgkin lymphoma or Hodgkin lymphoma) who have received any cytotoxic or radiation therapy
* Received treatment for leukemia or lymphoma 1-10 years ago

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Records from the practice of the study investigators will be reviewed to identify patients.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Quality of life | 1-10 years after treatment
Most common areas of concern | 1-10 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Regan Demshar, RN, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States